CLINICAL TRIAL: NCT03410550
Title: Exoskeleton Training After Spinal Cord Injury
Brief Title: Exoskeleton and Spinal Cord Injury
Acronym: EXTra-SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGuire Research Institute (Other)
Responsible Party: Principal Investigator, Ashraf Gorgey, Director of SCI Research, McGuire Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02375
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Twenty subjects will participate in a powered exoskeleton (EKSO) for one or twice a week for 12 weeks. The program will involve walking with the robotic suits for 1 hour for persons with complete (n=10) and persons with incomplete (n=10) SCI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exoskeleton Training (Experimental): Twenty men with complete and incomplete SCI will be enrolled in the trial.
  Interventions: Device: Exoskeleton Training

INTERVENTIONS:
Device: Exoskeleton Training — Twenty subjects will participate in a powered exoskeleton (EKSO) for one or twice a week for 12 weeks. The program will involve walking with the robotic suits for 1 hour for persons with complete (n=10) and persons with incomplete (n=10).

SUMMARY:
The purpose of the current study is to investigate the effects of powered exoskeleton (EKSO) on cardiovascular performance as measured by resting blood pressure and heart rate, peak oxygen consumption during walking, energy expenditure, whole and regional body composition assessments. The effects of exoskeleton training on walking kinematics including stand-up time, walking time, distance covered and speed of walking will also be evaluated.

DETAILED DESCRIPTION:
Powered exoskeletons using robotic suits have recently been introduced for the rehabilitation of persons with spinal cord injury (SCI). Exoskeletons offer a unique opportunity for persons with SCI to experience standing and walking at a low metabolic cost. Evidence suggested that exoskeleton assisted walking can decrease spasticity and improve bowel movement. Training may also improve the level of physical activity as well as psychological parameters that are likely to interfere with rehabilitation outcomes. Previous studies reported that a frequency of 2-3 times per week or more for 1-2 hours may be beneficial in the rehabilitation of persons with SCI. Using exoskeletal-assisted walking to improve the level of physical activity may be appealing to persons with SCI.

Exoskeleton training for 12 weeks may enhance energy expenditure, parameters of physical activity and result only on modest effects on both cardiovascular and body composition parameters. In other words, persons with tetraplegia may have greater cardiovascular and body composition adaptations compared to persons with paraplegia. Twenty subjects will participate in a powered exoskeleton (EKSO) for one or twice a week for 12 weeks. The program will involve walking with the robotic suits for 1 hour for persons with complete (n=10) and persons with incomplete (n=10) SCI.

ELIGIBILITY:
Inclusion Criteria:

1. A written clearance by the medical doctor .
2. Participants will have to be 1 year post-injury with any level of injury.
3. All participants will be between 18-70 years old, men/women,

Exclusion Criteria:

1. Participants with body weight greater than 220 lbs
2. Whole body T-scores less than -2.5 standard deviation will result in elimination from the program.
3. Hip width, upper leg length and lower leg length that do not fit in the robotic suit.
4. Previous unhealed fracture in both lower or upper extremities
5. Leg length discrepancy that is unlikely to be managed by having shoe inserts
6. High resting blood pressure greater than 130/80 mmHg
7. Sudden drop in blood pressure by 20 mmHg especially in persons with tetraplegia.
8. Medical conditions prior enrollment similar to cardiovascular disease, uncontrolled type II diabetes mellitus, uncontrolled hypertension, and those on insulin, pressures sores stage 2 or greater, or urinary tract infection or symptoms.
9. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (mmHg) | 12 weeks
  Resting blood pressure and post-exercise blood pressure will be measured every visit.
Walking time (minutes) | 12 weeks
  The robotic unit will measure standing up time, walking time and walking distance for every visit.
Oxygen uptake (l/min) | 12 weeks
  Oxygen uptake will be measured during sitting, standing and walking at the beginning and at the end of the training program.
Body Composition (kg) | 12 weeks
  Body composition using dual energy x-ray absorptiometry anthropometrics' will be measured during sitting, standing and walking at the beginning and at the end of the training program.

SECONDARY OUTCOMES:
Six minute-walk Test (meter) | 12 weeks
  The test will competed at the beginning and at the end of study to measure distance.
Walking Index for Spinal Cord Injury II (WISCI II) | 12 weeks
  The test will competed at the beginning and at the end of study
Electromyography (EMG) activity of 6 muscle groups (mV) | 12 weeks
  The test will competed at the beginning and at the end of study
Mitochondrial health using near infra-red spectroscopy (seconds) | 12 weeks
  The test will competed at the beginning and at the end of study
10 meter walk Test (m/sec) | 12 weeks
  The test will competed at the beginning and at the end of study to measure speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fresc.2021.789422/full